CLINICAL TRIAL: NCT00119145
Title: A Non-Inferiority, Open-Labelled, Randomised Trial Of The Efficacy And Safety Of Artesunate-Amodiaquine, Artemether-Lumefantrine, And Artesunate-Lapdap For Treatment Of Uncomplicated P. Falciparum Malaria Among Children In Ghana
Brief Title: Kintampo Trial of Combination Therapy for Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITDCVG44
Record Dates: First submitted 2005-07-04; First posted 2005-07-13 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: antimalarial drugs; efficacy; safety; trial
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: artesunate-amodiaquine
Drug: coartem
Drug: artesunate-lapdap

SUMMARY:
Case management is one of the key strategies for malaria control in most endemic countries. Plasmodium falciparum malaria is becoming resistant to commonly used and cheap antimalarial drugs such as chloroquine, amodiaquine, and sulfadoxine-pyrimethamine (SP). Thus the safety and efficacy of new anti-malarial drugs need to be tested in sites with well-characterised malariometric indices in order to make appropriate treatment policies.

Artemisinin-based combination chemotherapies have been documented to consistently produce faster relief of clinical symptoms and parasite clearance in uncomplicated falciparum malaria than any other currently used antimalarial drugs. So far, artesunate-amodiaquine (AS-AQ) and artemether-lumefantrine (AR-LM) are the only two registered fixed-dose artemisinin combination chemotherapies produced at industrial scale, with good manufacturing practices and already used in Africa. Several African countries, including Ghana, are therefore introducing either AS-AQ or AR-LM as first-line antimalarials or evaluating the case for such a change. Clearly, a direct comparison of both the safety and efficacy profiles of the two combinations under different epidemiological conditions is urgently needed to guide informed decisions on the most appropriate antimalarial first-line treatment regimen.

This study aims to evaluate the efficacy and safety of artesunate-amodiaquine combination therapy, artemether-lumefantrine, and artesunate-lapdap in an open-labelled, randomised, non-inferiority drug trial.

The study results will inform future decisions on first- and second-line treatments for uncomplicated P. falciparum malaria with respect to efficacy and safety in Ghana.

DETAILED DESCRIPTION:
A study funded by the GMP-LSHTM in the Kintampo district of Ghana is currently assessing the efficacy of SP as part of a comprehensive process of characterising the site into the patterns of seasonal dynamics of P. falciparum transmission, infection, and morbidity. The initial results from this study have demonstrated a high parasitological failure rate(18%) on day 14 of treatment, an indication that SP is no longer suitable for use in Ghana. Artesunate combination therapies (ACTs) have been found to be efficacious and safe, producing rapid clearance of parasites and malaria symptoms; they are very well tolerated. Lapdap is a newly registered, relatively cheap antimalarial with short half-life and has been found to be highly efficacious in strict trial conditions for treatment of acute uncomplicated falciparum infections in endemic sites in Africa. Despite the rapid clearance of lapdap, children treated with this drug did not have higher incidence of malaria episodes than those treated with SP though haematological adverse effects have been documented to be more common with lapdap than with SP. At present, the fixed-dose combination regimens of artesunate-amodiaquine (AS-AQ) and artemether-lumefantrine (AR-LM) are the only two registered artemisinin combination chemotherapies produced at industrial scale, with good manufacturing practices and already used in Africa. Several African countries are introducing either AS-AQ or AR-LM as first-line antimalarials or evaluating the case for such a change. Ghana, has just changed its antimalarial drug policy to artesunate-amodiaquine combination therapy (AS-AQ) as first line drug. The selection of this new ACT has been driven partly by cost of treatment, but a critical look at the safety and efficacy of ACTs in Ghana has yet to be done.

This study aims to evaluate the efficacy and safety of artesunate-amodiaquine combination therapy (AS-AQ), Artemether-lumefantrine (Coartem), and Artesunate-lapdap) in a drug non-inferiority study.

Objectives

Primary objective:

• To evaluate the efficacy of artesunate-amodiaquine versus artemether-lumefantrine, versus artesunate-lapdap in the treatment of children aged 6 months to ten years, infected with uncomplicated falciparum malaria, at the paediatric outpatient clinic in the Kintampo hospital.

Secondary objectives:

• To evaluate the safety of artesunate-amodiaquine versus artemether-lumefantrine, versus artesunate-lapdap in the treatment of children 6 months to ten years with uncomplicated falciparum malaria.

Study design and methods

Study site: This study is being conducted in Kintampo district in the middle belt of Ghana where the investigators in the Kintampo Health Research Centre are located. Kintampo Health Research Centre (KHRC), one of three research centres under the Health Research Unit (HRU) of the Ghana Health Service, Ghana, lies within the forest-savannah, transitional ecological zone in the Brong Ahafo Region of Ghana.

Study design:

This is a randomised, open-labelled, non-inferiority drug trial. At the Kintampo district hospital, 510 paediatric outpatients (refer sample size calculation) with uncomplicated P. falciparum malaria and aged between 6 months and 10 years will be recruited and randomly assigned to one of the three study arms: (i) Artesunate-Amodiaquine (AS-AQ), (ii) Artemether-Lumefantrine (AR-LM), or (iii) Artesunate-lapdap (AS-LP). The classification of clinical and parasitological responses will follow the relevant WHO protocol for areas of intense transmission. Follow-up, however, will be extended beyond day 14 up to day 28 to increase the sensitivity of the in vivo test. PCR-based genotyping comparing pairs of parasite isolates from day 0 and day of asexual parasite reappearance will be used to distinguish between recrudescence and re-infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 10 years
* Body weight >5 kg
* Uncomplicated P. falciparum malaria
* Mono-infection with P. falciparum
* Asexual parasite density 2,000 to 200,000 parasites/µl
* Haemoglobin ≥7.0 g/dL
* Axillary temperature ≥37.5ºC or history of fever in preceding 24 hr
* Ability to tolerate oral therapy
* Residence in study area

Exclusion Criteria:

* Haemoglobin <7.0 g/dL
* Leucocyte count: >15,000/µL
* G6PD deficiency
* Mixed malaria infections
* Danger signs (unable to drink; repeated vomiting; recent history of convulsions; lethargic or unconscious state; unable to stand up or to sit) and signs of severe malaria as defined by WHO
* Any other severe underlying disease (cardiac, renal, hepatic diseases, malnutrition, known HIV infection)
* Concomitant disease masking assessment of response, e.g. known or suspected hearing impairments

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 510 (Estimated)
Dates: Start 2005-06; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
adequate clinical and Parasitological response (ACPR)by day 28.

SECONDARY OUTCOMES:
Parasitological cure rate by day 14
Parasitological cure rate by day 28
Clinical cure rates by days 14 and 28
Incidence rates of adverse events
Gametocyte carriage at days 7, 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Seth Owusu-Agyei, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, MBBS, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Brian M Greenwood, FRCP, FRS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Kintampo Health Research Centre, Kintampo, Brong Ahafo Region, Ghana

REFERENCES:
- [Derived] Owusu-Agyei S, Asante KP, Owusu R, Adjuik M, Amenga-Etego S, Dosoo DK, Gyapong J, Greenwood B, Chandramohan D. An open label, randomised trial of artesunate+amodiaquine, artesunate+chlorproguanil-dapsone and artemether-lumefantrine for the treatment of uncomplicated malaria. PLoS One. 2008 Jun 25;3(6):e2530. doi: 10.1371/journal.pone.0002530. PMID 18575626